CLINICAL TRIAL: NCT01054872
Title: A Phase 1B Clinical Trial to Examine the Role of Host Genetics in Determining the Immune Response to HIV Vaccination (With VRC-HIVDNA016-00-VP and VRC-HIVADV014-00-VP) in Twin Pairs
Brief Title: Examining the Role of Genetics in Determining the Immune Response to an HIV Vaccine in HIV-Uninfected Adult Twins
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: HVTN 082; 10771 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 2010-01-21; First posted 2010-01-22 (Estimated); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: HIV Seronegativity; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Monozygotic (MZ) Twins (Experimental): Participants will receive the DNA vaccine at baseline and Months 1 and 2. They will then receive the rAd5 vaccine at Month 6.
  Interventions: Biological: HIV-1 DNA plasmid vaccine; Biological: HIV-1 recombinant Ad5 vaccine
- Dizygotic (DZ) Twins (Experimental): Participants will receive the DNA vaccine at baseline and Months 1 and 2. They will then receive the rAd5 vaccine at Month 6.
  Interventions: Biological: HIV-1 DNA plasmid vaccine; Biological: HIV-1 recombinant Ad5 vaccine

INTERVENTIONS:
Biological: HIV-1 DNA plasmid vaccine — 4 mg injection administered as 1 mL intramuscularly via Biojector in deltoid
  Other Names: VRC-HIVDNA016-00-VP
Biological: HIV-1 recombinant Ad5 vaccine — 1 x 10^10 particle units (PU) administered as 1 mL intramuscularly by needle and syringe in deltoid
  Other Names: VRC-HIVADV014-00-VP

SUMMARY:
The purpose of this study is to examine the role of genetics in determining the immune response to an HIV vaccine in pairs of HIV-uninfected twins.

DETAILED DESCRIPTION:
Genetics may play a role in the immune response to HIV vaccines. It remains unknown, however, exactly what the genetic influence on the immune response may be. This study will examine how genes affect the strength of an immune response produced by HIV vaccines and how genes influence different immune responses. In this study, participants will receive two HIV vaccines-a DNA HIV vaccine (VRC-HIVDNA016-00-VP) and a recombinant adenoviral serotype 5 (rAd5) vector HIV vaccine (HIVADV014-00-VP). Both of these vaccines are experimental, but have been used in previous clinical trials without any serious side effects. Comparing immunological responses in HIV vaccine trials can be complicated by various genetic and environmental factors. This study will enroll pairs of twins who grew up in common childhood environments. This will provide researchers with participants who have similar backgrounds so that the role of genetics can be examined while controlling for other environmental variables. The purpose of this study is to examine how genes may influence the immune response to a DNA HIV vaccine followed by a rAd5 HIV vaccine.

This study will enroll pairs of healthy, HIV-uninfected monozygotic and dizygotic adult twins. Participants will receive the DNA vaccine at baseline and Months 1 and 2, and the rAd5 vaccine at Month 6. Both vaccines will be injected into the upper arm. At all vaccination study visits, participants will undergo a medical history and medication history review, physical exam, and blood collection. Participants will also complete questionnaires and a social impact assessment. They will receive counseling on HIV testing, risk reduction, and pregnancy prevention. After receiving the vaccine, participants will remain in the clinic for at least 30 minutes for observation and monitoring of side effects. For 3 days after each vaccination, participants will record their temperature and side effects in a symptom log. In addition to the vaccine study visits, additional study visits will occur at Weeks 2, 6, and 10; 1, 3, and 7 days after the Month 6 visit; and Months 7, 9, 12, and 18. Various study procedures, including a physical exam, blood collection, and counseling, will be repeated at these visits. At the end of 18 months, participants will be contacted by study researchers once a year for 3 ½ years for follow-up health monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Pairs of MZ and DZ twins who shared common childhood environments
* If born male, participant must be fully circumcised (as documented at screening examination). Circumcision must have been performed at least 90 days prior to first vaccination and surgical site must be fully healed.
* Access to a participating HIV Vaccine Trials Network (HVTN) clinical research site (CRS) and willing to be followed for the duration of the study
* Assessment of understanding, including the completion of a questionnaire before the first vaccination and demonstration of understanding for all questionnaire items answered incorrectly
* Willing to receive HIV test results
* Willing to discuss HIV infection risks, amenable to HIV risk reduction counseling, committed to maintaining behavior consistent with low risk HIV exposure through the last required study visit, and willing to continue annual follow-up contact after the final study visit for a total of 5 years after study entry
* In good general health, as shown by medical history, physical exam, and screening laboratory tests
* Assessed by the clinic staff as having a "low risk" for HIV infection on the basis of sexual behaviors in the 12 months before study entry. More information on this criterion can be found in the protocol.
* Ad5 nAb titer less than 1:18
* Hemoglobin greater than or equal to 11.3 g/dL for participants who were born female, and greater than or equal to 13.0 g/dL for participants who were born male
* White blood cell count between 3,300 to 12,000 cells/mm^3
* Total lymphocyte count greater than or equal to 800 cells/mm^3
* Remaining differential either within site's normal range or with site physician approval
* Platelet level between 125,000 to 550,000/mm^3
* Alanine aminotransferase (ALT) less than or equal to 2.5 times the site's upper limit of normal
* Negative HIV-1 and -2 blood test
* Negative Hepatitis B surface antigen (HBsAg)
* Negative anti-Hepatitis C virus antibodies (anti-HCV), or negative HCV polymerase chain reaction (PCR) if the anti-HCV test is positive
* Participants who were born female must have a negative pregnancy test result before the first study vaccination
* Agree not to participate in any other study requiring blood draws more than 10 mLs total or additional investigational drugs 56 days before study entry or during the study
* Participants who were born female must agree to use an effective form of contraception from at least 21 days before study entry until the last study visit. More information on this criterion can be found in the protocol.
* Participants who were born female must agree not to seek pregnancy through alternative methods (e.g., artificial insemination, in vitro fertilization) until after the last study visit

Exclusion Criteria:

* Excessive daily alcohol use, frequent binge drinking, chronic marijuana abuse, or use of any other illicit drugs in the 12 months before study entry
* History of newly acquired syphilis, gonorrhea, non-gonococcal urethritis, herpes simplex virus type 2, chlamydia, pelvic inflammatory disease (PID), trichomonas, mucopurulent cervicitis, epididymitis, proctitis, lymphogranuloma venereum, chancroid, or hepatitis B in the 12 months before study entry
* Received HIV vaccines in a prior HIV vaccine trial
* Immunosuppressive medications received within 168 days before the first study vaccination
* Blood products received within 120 days before the first study vaccination
* Immunoglobulin received within 60 days before the first study vaccination
* Live attenuated vaccines received within 30 days before the first study vaccination or scheduled within 14 days after injection
* Investigational research agents received within 30 days before the first study vaccination
* Intent to participate in another investigational drug study
* Any vaccines that are not live attenuated vaccines or allergy treatment with antigen injections received within 14 days before the first study vaccination
* Current anti-tuberculosis preventive therapy or treatment
* Clinically significant medical condition, abnormal physical examination findings, abnormal laboratory results, or past medical history that may affect current health
* Any medical, psychiatric, occupational, or other condition that would interfere with participation in the study
* Serious adverse reactions to vaccines, including anaphylaxis and related symptoms (e.g., hives, respiratory difficulty, angioedema, abdominal pain). A person who had an adverse reaction to the pertussis vaccine as a child is not excluded.
* Autoimmune disease or immunodeficiency
* Active syphilis infection
* Asthma, other than mild, well-controlled asthma. More information on this criterion can be found in the protocol.
* Type 1 or type 2 diabetes mellitus, including cases controlled with diet alone. People with a history of isolated gestational diabetes are not excluded.
* Surgical removal of the thyroid or thyroid disease requiring medication during the 12 months before study entry
* History of hereditary angioedema, acquired angioedema, or idiopathic forms of angioedema
* Idiopathic urticaria within the 2 years before study entry
* High blood pressure that is not well controlled OR blood pressure of 150/100 mm Hg or greater at study entry. More information on this criterion can be found in the protocol.
* Bleeding disorder (e.g., factor deficiency, coagulopathy, platelet disorder requiring special precautions)
* Cancer. People with surgically removed cancer that, in the opinion of the investigator, is unlikely to recur are not excluded.
* Seizure disorder. People with a history of seizures who have not required medications or had a seizure within the 3 years before study entry are not excluded.
* Absence of the spleen
* Psychiatric condition that makes study compliance difficult (e.g., people with psychoses in the 3 years before study entry, ongoing risk for suicide, history of suicide attempt in the 3 years before study entry)
* Pregnant or breastfeeding

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2010-01; Primary Completion 2012-11 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Magnitude of HIV-1 insert-specific cellular responses, as measured by ELISpot, intracellular cytokine staining (ICS), or other modalities | Measured at 4 weeks after the rAd5 boost
Magnitude of Ad-specific cellular responses, as measured by ELISpot, ICS, or other modalities | Measured at 4 weeks after the rAd5 boost

SECONDARY OUTCOMES:
Number of HIV epitopes targeted by CD4 and CD8 T-cells, as measured by ELISpot, ICS, or other modalities | Measured at 4 weeks after the rAd5 boost
Number of Ad epitopes targeted by CD4 and CD8 T-cells, as measured by ELISpot, ICS, or other modalities | Measured at 4 weeks after the rAd5 boost
Percentage of insert-specific T lymphocytes expressing 1, 2, or 3 cytokines, as measured by HIV-1 specific multi-parameter ICS or other modalities | Measured at 4 weeks after the rAd5 boost
Percentage of Ad-specific T lymphocytes expressing 1, 2, or 3 cytokines, as measured by HIV-1 specific multi-parameter ICS or other modalities | Measured at 4 weeks after the rAd5 boost
HIV-1-specific nAb titers, as measured by antibody titer assays | Measured at 4 weeks after the rAd5 boost
Ad-specific nAb titers, as measured by antibody titer assays | Measured at 4 weeks after the rAd5 boost
Serum concentration of IL-6, IL 12, TNF-a, INF-y, IL-1Ra, IP-10/CXCL-10, and MCP-1/CCL2 (and other circulating cytokines associated with the innate immune response, as measured by Luminex assay or other modality) | Measured at baseline, and Days 0, 1, 3, and 7 after the rAd5 boost
Numbers of circulating peripheral blood lymphocytes, monocytes, and neutrophils | Measured at baseline, and Days 0, 1, 3, and 7 after the rAd5 boost
Local and systemic reactogenicity signs and symptoms, laboratory measures of safety, adverse events (AEs), and AEs reported on an expedited basis to DAIDS (EAEs) | Measured throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Baden, Study Chair — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Brigham and Women's Hospital Vaccine CRS (BWH VCRS), Boston, Massachusetts
  - Seattle Vaccine and Prevention CRS, Seattle, Washington

REFERENCES:
- [Background] Hunt PW, Carrington M. Host genetic determinants of HIV pathogenesis: an immunologic perspective. Curr Opin HIV AIDS. 2008 May;3(3):342-8. doi: 10.1097/COH.0b013e3282fbaa92. PMID 19372988
- [Background] Newport MJ, Goetghebuer T, Marchant A. Hunting for immune response regulatory genes: vaccination studies in infant twins. Expert Rev Vaccines. 2005 Oct;4(5):739-46. doi: 10.1586/14760584.4.5.739. PMID 16221074